CLINICAL TRIAL: NCT06607159
Title: Childhood Obesity Prevention Project in Gran Canaria
Acronym: POI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Complejo Hospitalario Universitario Insular Materno Infantil (Other)
Collaborators: FundaciÃ³n Canaria de InvestigaciÃ³n Sanitaria (Unknown); Instituto Universitario de Investigaciones BiomÃ©dicas y Sanitarias (iUIBS) de la Universidad de Las (Unknown)
Responsible Party: Principal Investigator, Yeray Nóvoa Medina, Principal Investigator, Complejo Hospitalario Universitario Insular Materno Infantil
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2020-356-1
Record Dates: First submitted 2024-09-12; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Weight Change; BMI; Activity Level; Cholesterol (total and HDL); Glucose; Body Composition Changes
Keywords: children; obesity prevention; schools; multicomponent
MeSH Terms: conditions — Body Weight Changes

STUDY DESIGN:
Intervention Model Description: This is a cluster-randomized, controlled, parallel clinical trial assessing the impact of an educational intervention in the prevalence of obesity in children. The inclusion in both arms of the study was randomized with a 1:1 ratio (even though we performed cluster randomization, the aim was to have a 1:1 participants´ratio, not a 1:1 classroom ratio). To randomize the participant schools, we employed a stratified cluster randomization approach. First, we categorized schools into three types: public, private, and subsidized. Within each category, we assigned a random number to each school a and then ranked them from highest to lowest based on these numbers. Given that we knew the number of children in each class, we started allocating schools with the highest random numbers to either the intervention or control arm, continuing this process until the target number of children in each arm was reached. All children from a given school were assigned to the same study arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Group of children in whom the protocol is implemented (the whole class)
  Interventions: Other: Implementation of healthy habits teaching protocol
- Control (No Intervention): Group of children in whom the protocol is not implemented (the whole class)

INTERVENTIONS:
Other: Implementation of healthy habits teaching protocol — Protocol for teaching healthy lifestyle habits, aimed at school-age children (initially between 1st and 4th grade of primary school), to be implemented transversally in schools. This protocol takes into account three levels of action: school, family and pupils. It includes materials in paper format and digital materials, that can be used both at school and at home.
  Arms: Intervention

SUMMARY:
Given the alarming rates of obesity and overweight in our child population, the investigators have developed an intervention strategy, based on a multidisciplinary, school-centered approach, which addresses nutritional education, physical activity, behavioral intervention techniques and tools that facilitate the learning of healthy lifestyle habits in children between 6 and 10 years of age.

DETAILED DESCRIPTION:
This is a cluster-randomized, controlled, parallel clinical trial assessing the impact of an educational intervention in the prevalence of obesity in children.

Boys and girls aged 6-10 years (1st to 4th grades of primary school) from public, state-subsidized and private schools on the island of Gran Canaria, Canary Islands, Spain, were recruited. The selection of schools was based on convenience. After obtaining a list of schools from contacts with the local diabetic association and members of the team, the project was explained and schools were invited to participate. After obtaining the consent from several schools, the inclusion in both arms of the study was randomized with a 1:1 ratio (even though we performed cluster randomization, the aim was to have a 1:1 participants´ratio, not a 1:1 classroom ratio), and the parents of the students in the aforementioned classes were invited to participate. Finally, those children whose parents consented to their participation were included. To randomize the participant schools, the researchers employed a stratified cluster randomization approach. First, the researchers categorized schools into three types: public, private, and subsidized. Within each category, the researchers assigned a random number to each school and then ranked them from highest to lowest based on these numbers. Given that the researchers knew the number of children in each class, the researchers started allocating schools with the highest random numbers to either the intervention or control arm, continuing this process until the target number of children in each arm was reached. This approach ensured a 1:1 ratio of participants between arms while maintaining randomization integrity, even though it could result in an unequal number of schools per arm. To maintain cluster integrity, all children from a given school were assigned to the same study arm. Randomization was performed by the main investigator (YNM). No changes to the methodology were implemented after trial commencement.

The project for the prevention of childhood obesity in the Canary Islands seeks to increase knowledge about healthy lifestyle habits in the pediatric age group as a tool to reduce the rate of childhood overweight and obesity (based on recommendations on diet, physical activity, leisure time devoted to screens and hours of sleep published by official bodies such as the WHO, the American Academy of Pediatrics (AAP) and the American Centre for Disease Control and Prevention (CDC)). One of the main goals of the research team was to develop cost-free strategies and tools for schools. To achieve this, the researchers decided to involve teachers as the primary drivers of change and schools as the implementation sites for the study protocol. To this end, the pediatric endocrinology and gastroenterology units of the Complejo Hospitalario Universitario Materno Infantil de Las Palmas de Gran Canaria have collaborated with the group specializing in Learning Difficulties, Psycholinguistics and Information and Communication Technologies; of the University of La Laguna (https://viinv.ull.es/grupos/1119/), which includes psychologists, teachers and pedagogues among its members.

As a result of this collaboration, a protocol for teaching healthy lifestyle habits has been developed, aimed at school-age children (initially between 1st and 4th grade of primary school), to be implemented transversally in schools. This protocol takes into account three levels of action: school, family and pupils.

1. Materials in paper format: These materials are mainly used in the classroom, although they can also be used at home. They have been designed according to the grade level and the level of competence of the students. These workbooks are based on the curricular contents linked to healthy lifestyle habits that should be worked on according to the school year as established in DECREE 89/2014, of 1 August, which establishes the organization and curriculum of Primary Education in the Autonomous Community of the Canary Islands (19). Likewise, from an inclusive perspective, suitable materials have been designed for students with Specific Educational Support Needs (SEN) that make it difficult for them to access the written code (Image 1a). The books can be found in the following link: https://www.fundacionmapfrecanarias.org/formacion-prevencion/actividades-didacticas/programa-obesidad-infantil-fmc/
2. Digital materials: Gamification has been proven to motivate and promote improvements in the nutrition of children(20). For our intervention, 6 games have been designed in application format aimed at increasing daily physical activity time (2 games: 5 minutes of movement and active breaks), a balanced diet (2 games: healthy breakfasts and the cool recipe) and knowledge and reflection on healthy lifestyle habits (2 games: asking questions and my alien) (Image 1b). The digital materials are embedded in a web platform that allows teachers to know the health status of the classroom based on the scores obtained by the students in each of the mini-games. The games can be used in the classroom or at home (with a time limit of 30 min/day), thus trying to facilitate parental interaction with the program. It is important to emphasize that we will always work with the classroom score, emphasizing that health is everyone´s responsibility.

The project has an evaluation phase (April-June 2022), a teacher training phase (April-June 22) and a teaching project implementation phase (school year 2022-2023).

ELIGIBILITY:
Inclusion Criteria:

* Children between 6-10 years of age, studying in the recruited schools, who consented to participate in the study

Exclusion Criteria:

* Children younger than 6 or older than 10 years of age, who did not conset to participate in the study

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 557 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Changes in body mass index from baseline to post-intervention in the control group vs the intervention group | 1 year
  Body mass index (weight in kg/height in meters squared) will be determined after weight and height have been measured both at baseline and after the intervention period. The change in BMI from the control and intervention groups will be compared to determine if there is a difference in the rate of change between both groups.

SECONDARY OUTCOMES:
Changes in percentage of body fat between the control and intervention group, measured with an impedance scale | 1 year
  The investigators will determine de percentage of body fat using the Tanita Impedance Scale (Tokyo, Japan) model DC-360. The rate of change in the percentage of body fat between the 2 groups will be compared at the end of the study period.
Changes in weight from baseline to post-intervention in the control group vs the intervention group | 1 year
  The investigators will determine de weight of all children using the Tanita Impedance Scale (Tokyo, Japan) model DC-360. The rate of change between the 2 groups will be compared at the end of the study period.
Changes in waist circumference between the control and intervention group, measured with an anthropometric flexible, non-stretchable measuring tape | 1 year
  The investigators will determine de waist circumference of all children using an anthropometric flexible, non-stretchable measuring tape. The rate of change between the 2 groups will be compared at the end of the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Yeray Nóvoa, MD, MPH, PhD, Principal Investigator — Instituto Universitario de Investigaciones Biomédicas y Sanitarias (iUIBS) de la Universidad de Las
Locations (1):
- CHUIMI, Las Palmas de Gran Canaria, Canary Islands, Spain

IPD SHARING:
Plan to Share IPD: No
there is no need to share IPD data

REFERENCES:
- See also: Link that describes the study, as well as shares the printed material used by the teachers — https://www.fundacionmapfrecanarias.org/formacion-prevencion/actividades-didacticas/programa-obesidad-infantil-fmc/